CLINICAL TRIAL: NCT02073643
Title: Delay Discounting and Household Food Choices
Brief Title: Study of Household Purchasing Patterns, Eating and Recreation
Acronym: SHoPPER
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Collaborators: University of Minnesota (Other); University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Brad Appelhans, Assistant Professor of Preventive Medicine, Rush University Medical Center
Other Study IDs: 12051001
Record Dates: First submitted 2014-02-24; First posted 2014-02-27 (Estimated); Results first posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Dietary Habits; Adiposity; Blood Pressure
MeSH Terms: conditions — Feeding Behavior; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This project examines behavioral and household characteristics associated with food purchasing patterns.

ELIGIBILITY:
Inclusion Criteria:

1. Adult individual who reports making at least 75% of household food purchases
2. Resides in City of Chicago, Illinois or surrounding suburbs

Exclusion Criteria:

1. Inability to provide informed consent in English
2. Living in transitional housing or on a college campus
3. Lack of a cellular or land line phone
4. Gang presence or illegal activity in the immediate vicinity of the home, or other factors jeopardizing researcher safety during home visits (e.g., extreme unsanitary conditions)
5. Having a household member, including the primary shopper, with a medical condition or food allergy that substantially influences household food choices (e.g., phenylketonuria, celiac disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chicago households
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2013-11; Primary Completion 2016-11 (Actual); Study Completion 2018-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Appelhans BM, Tangney CC, French SA, Crane MM, Wang Y. Delay discounting and household food purchasing decisions: The SHoPPER study. Health Psychol. 2019 Apr;38(4):334-342. doi: 10.1037/hea0000727. PMID 30896220
- [Derived] French SA, Tangney CC, Crane MM, Wang Y, Appelhans BM. Nutrition quality of food purchases varies by household income: the SHoPPER study. BMC Public Health. 2019 Feb 26;19(1):231. doi: 10.1186/s12889-019-6546-2. PMID 30808311
- [Derived] Appelhans BM, French SA, Tangney CC, Powell LM, Wang Y. To what extent do food purchases reflect shoppers' diet quality and nutrient intake? Int J Behav Nutr Phys Act. 2017 Apr 11;14(1):46. doi: 10.1186/s12966-017-0502-2. PMID 28399887

RESULTS

PARTICIPANT FLOW:
Groups:
- Main Food Purchasing Cohort: This is a cohort study.
Period: Overall Study
Arm/Group | Main Food Purchasing Cohort
Started | 204
Completed | 180
Not Completed | 24
Not completed — Lost to Follow-up | 24

BASELINE CHARACTERISTICS:
Groups:
- Main Cohort: This is a cohort study.
Arm/Group | Main Cohort
Number analyzed (Participants) | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.11 (13.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169
  Male | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 93
  White | 73
  More than one race | 27
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 204
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 31.15 (9.08)
Delay discounting [Mean (Standard Deviation); unit: (Value of $100) * (days until receipt)] — Area under the curve of delay discounting indifference points for hypothetical monetary rewards, on scale from 0-100.
  (Value of $100) * (days until receipt) | 32.77 (28.54)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg, systolic] — Systolic blood pressure taken in triplicate, at rest in seated position.
  mmHg, systolic | 120.19 (15.29)

OUTCOME MEASURES:

1. Primary Outcome: Diet Quality of Household Food Purchases
Description: Diet quality was quantified by applying the Healthy Eating Index-2015 (HEI-2015) scoring criteria (https://epi.grants.cancer.gov/hei/) to the nutrient and food group data of purchased foods and beverages. The HEI-2015 scores adherence to the Department of Health and Human Services' 2015 Dietary Guidelines for Americans. Adherence to recommended intakes for 13 key dietary components is scored on continuous scale for each component, and the 13 component scores are then summed to obtain a total score ranging from 0-100. Higher scores reflect closer adherence to the dietary guidelines.
Time Frame: 2 weeks
Population: N=202 participants had food purchase data available for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Main Cohort
Number analyzed (Participants) | 202
units on a scale | 57.88 (15.22)

2. Secondary Outcome: Diet Quality of Dietary Intake
Description: Diet quality was quantified by applying the Healthy Eating Index-2015 (HEI-2015) scoring criteria (https://epi.grants.cancer.gov/hei/) to the nutrient and food group data derived from three 24-hour diet recalls. The HEI-2015 scores adherence to the Department of Health and Human Services' 2015 Dietary Guidelines for Americans. Adherence to recommended intakes for 13 key dietary components is scored on continuous scale for each component, and the 13 component scores are then summed to obtain a total score ranging from 0-100. Higher scores reflect closer adherence to the dietary guidelines.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Main Cohort
Number analyzed (Participants) | 204
units on a scale | 59.49 (14.38)

3. Secondary Outcome: Home Food Environment
Description: Availability of obesity promoting foods in the home, assessed with an audit-based inventory. The audit captures the presence of 71 "obesity promoting" foods. The sum of these items ranges from 0-71, with higher scores reflecting greater availability in the home.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Main Cohort
Number analyzed (Participants) | 204
units on a scale | 20.19 (8.76)

4. Secondary Outcome: Percentage of Total Energy Purchased From Non-store Sources (e.g., Fast Food and Take-out/Delivery, Restaurants)
Description: Percentage of total energy (kcal) purchased from all sources other than food stores/supermarkets, including fast food and take-out/delivery, full-service restaurants, vending machines, bars/taverns, and cafeterias.
Time Frame: 2 weeks
Population: N=202 subjects had food purchase data available for analysis
Measure: Median (Inter-Quartile Range); unit: Percentage of total energy purchased
Arm/Group | Main Cohort
Number analyzed (Participants) | 202
Percentage of total energy purchased | 10.65 [2.55 to 24.01]

5. Other Pre Specified Outcome: Change From Baseline in Systolic Blood Pressure at 12 Months
Description: Change in systolic blood pressure
Time Frame: 12 months
Population: N=179 participants had blood pressure readings at both baseline and the 12-month follow up.
Measure: Mean (Standard Deviation); unit: change in mmHg, systolic
Arm/Group | Main Cohort
Number analyzed (Participants) | 179
change in mmHg, systolic | 1.00 (14.02)

6. Other Pre Specified Outcome: Change From Baseline in Body Mass Index at 12 Months
Description: Change in body mass index over 12 months of follow up
Time Frame: 12 months
Population: N=180 participants completed the 12-month follow up assessment
Measure: Mean (Standard Deviation); unit: difference in kg/m^2
Arm/Group | Main Cohort
Number analyzed (Participants) | 180
difference in kg/m^2 | 0.23 (1.69)

ADVERSE EVENTS:
Description: As this was an observational study, adverse events were not defined in advance. All-cause mortality, serious, and other adverse events were not monitored.
Arm/Group | Main Cohort
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No